CLINICAL TRIAL: NCT06432114
Title: Coping Through Sensory Modulation. A Sensory Awareness Program (SAP) for Reducing Anxiety and Mobilizing Coping Strategies for People With Severe Mental Health Problems. A Randomized Controlled Trial.
Brief Title: Sensory Awareness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAP
Record Dates: First submitted 2024-04-17; First posted 2024-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Awareness Program (Experimental)
  Interventions: Behavioral: Sensory Awareness Program (SAP); Other: Treatment as usual (TAU)
- Treatment as usual (Other)
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Sensory Awareness Program (SAP) — SAP is a new rehabilitation program for people with severe mental health problems. SAP aims to help the target group manage anxiety outburst and live an active life through sensory modulation techniques.
  Arms: Sensory Awareness Program
Other: Treatment as usual (TAU) — Treatment as usual is standard psychiatric care for the target group.

SUMMARY:
Few alternatives to addictive medical treatment exists for persons with severe mental health problems (SMHP) and anxiety, often connected to high risk of suicide. Access to effective interventions that depart in individuals' needs to cope with anxiety in everyday life is crucial to provide and desperately warranted by service users. Service users are often unaware of sensory needs, connected to anxiety outburst. The Sensory Awareness Program (SAP) is a group-based self-management intervention of 10 weeks developed to meet complex needs of regulating anxiety and related self-destructive behaviors. SAP stems from theories on sensory modulation and is an approach to manage physiological arousal associated with anxiety through self-regulated sensory-based coping strategies. International research show that sensory modulation is effective both as a method to reduce anxiety and thus restraint in acute mental health services (MHS), and also to empower users. However, much research to date focus on using sensory strategies within wards. International research and pre-studies of testing the SAP in outpatient MHS indicate that it is a promising self-management intervention to support everyday life. Earlier studies further show that users' unawareness of sensory needs triggers anxiety, and that anxiety itself is the main contributing factor for disrupting everyday life. Also, staff acknowledge sensory modulation but lack knowledge on whether programs such as SAP is effective and possible to implement.

The overall aim is to investigate the effectiveness of SAP as compared to treatment as usual (TAU) among 200 outpatients. The investigators hypothesize that SAP will be more effective than TAU in terms of reduced anxiety (primary outcome) at three months follow-up. Secondary clinical and personal recovery outcomes post intervention and at three and six months follow up will also be targeted and assumed to be in favour of the SAP group. The implementation process of the SAP will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Be assigned to a MHS
* Age over 18
* Having SMHP (including a diagnosis of mood disorder, anxiety disorder, eg PTSD, panic disorder etc, and/or psychotic disorder)
* Experience anxiety

Exclusion Criteria:

* Acutely mentally unwell
* Cognitively impaired
* Non-Swedish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, non-binary
Enrollment: 207 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Becks anxiety inventory (BAI) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire measuring the severity of anxiety symptoms with 21 questions, each describing a symptom of anxiety. The participant rates each item on a scale from 0 to 3, indicating how much he/she experiences each symptom. The scores range from 0 to 63, with higher scores indicating more severe levels of anxiety.

SECONDARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Hopkins Symptoms Checklist (HSCL-25) is a widely used screening instrument with 25 items measuring symptoms of anxiety and depression. The scale for each question includes four response categories from 1 (not at all) to 4 (very much). The total score is the average of all 25 items.
Difficulties in Emotion Regulation scale (DERS) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Difficulties in Emotion Regulation Scale (DERS) is a self-report measure of emotion regulation difficulties. The total score ranges from 16-80 with higher scores indicating more difficulties with emotion regulation.
Coping Orientation of Problem Experience Inventory (COPE) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Brief-COPE is an instrument reflecting individuals' coping strategies when exposed to a stressful situation. Brief-COPE is the short version and consists of 14 sub-scales, with 2 items in each scale, with a total of 28 items. The items are rated on a scale from 1 (seldom) to 4 (very often). In the current study, we will use the three-factor model of the instrument where the 14 subscales are divided into 3 factors; 'Problem-focused coping', 'Emotion-focused coping' and 'Avoidant coping'.
Manchester Short Assessment of Quality of Life Scale (MANSA) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Manchester Short Assessment of Quality of Life (MANSA) consists of 16 questions, covering different domains of life such as physical health, social relationships, employment, and overall life satisfaction. Each question is rated on a scale from 1 to 7, with higher scores indicating better quality of life.
Pearlin Mastery Scale | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Pearlin Mastery Scale is used to assess an individual's perceived sense of control over their life circumstances, containing seven questions to rate the level of agreement with statements about the ability to control and influence life. It covers areas such as personal growth, problem-solving, and self-mastery and is rated on a scale from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating greater levels of mastery.
Process of Recovery Questionnaire (QPR-7) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The Process of Recovery Questionnaire (QPR-7) is a short version of the instrument with 15 items (Argentzell et al., 2017). QPR-7 has seven questions concerning which aspects of recovery have been meaningful for the participants on a five-graded scale from 0 (disagree strongly) to 4 (agree strongly).
Profiles of Occupationa Engagement (POES) | Before intervention, post intervention (at 3 months), 6 and 9 months
  POES is an instrument that helps to discern the level of occupational engagement. The POES has two parts, one being the 24-hour yesterday time use diary and a second part consisting of a self-rated questionnaire with 9 items representing different components of occupational engagement. Based on the time diary the participants reflect on the content and rate to what extent it corresponds to a lower or higher level of occupational engagement on a 4-point scale.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Before intervention, post intervention (at 3 months), 6 and 9 months
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) is a questionnaire used to assess an individual's perceived level of functioning and disability across six domains of life with 12 questions covering: activities and participation in society. Each question is rated on a scale from 0 to 4, with higher scores reflecting greater levels of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skåne, Helsingborg, Sweden

REFERENCES:
- [Derived] Forsberg K, Sutton D, Stjernsward S, Bejerholm U, Argentzell E. Implementation of a sensory modulation intervention in mental health outpatient services: a process evaluation study. BMC Psychiatry. 2025 Jun 5;25(1):581. doi: 10.1186/s12888-025-07034-5. PMID 40474152